CLINICAL TRIAL: NCT04373421
Title: Effect of St. John's Wort Oil and Olive Oil on the Postoperative Complications After Impacted Third Molar Surgery: Randomized, Double-blind Clinical Trial
Brief Title: Effect of St. John's Wort and Olive Oils on the Postoperative Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01.08.2018/08
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — chlorhexidine gluconate; Mouthwashes; Benzydamine; Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- chlorhexidine gluconate plus benzydamine hydrochloride (Active Comparator): Chlorhexidine is one of the most commonly used medications after tooth extraction. It exhibits a wide spectrum of antiseptic, bactericidal and bacteriostatic effects. The most common side effect of chlorhexidine is oral discoloration, taste changes and allergic responses. Furthermore, it has been reported that chlorhexidine has cytotoxic effect on gingival fibroblasts, epithelial cells, neutrophils and red blood cells; also shows incremental trend in genotoxicity as the duration of usage is increased. Benzydamine hydrochloride is a nonsteroidal anti-inflammatory drug that elicits anti-inflammatory, analgesic, anesthetic and antimicrobial effects. It is often used in addition to the topical application of chlorhexidine.. However, side effects such as urticaria, erythema, pruritus, photosensitivity, bronchospasm and renal problems can be observed associated with the use of benzydamine.
  Interventions: Drug: Chlorhexidine Gluconate 0.12 % Mouthwash + benzydamine hydrochloride
- St. John's wort oil (Active Comparator): St. John's Wort (Hypericum perforatum) is a European medicinal plant with a history of more than 2000 years which possessing a variety of important constituents including phloroglucinols (hyperforin and adhyperforin), naphthodianthrones (hypericin and pseudohypericin), xanthones, essential oil, biflavones (biapigenin and amentoflavone), flavonol derivatives and phenolic compounds. The important components of St. John's Wort such as hypericin and hyperforin exert anti-inflammatory, antimicrobial, anticancer effects as well as stimulating tissue growth and differentiation. Hypericin exhibits anti-inflammatory effects by inhibiting the production of interleukin-12; whereas hyperforin reveals this effect by inhibiting the mechanisms of cyclooxygenase 1, 5-lipoxygenase and prostaglandin E2. St. John's Wort oil is extracted by maceration of the hypericum herb in carrier oil, such as virgin olive oil.
  Interventions: Procedure: St. John's wort oil
- Virgin olive oil (Active Comparator): The olive oil, a product extracted from the fruit of Olea europaea, exerts also antioxidant and anti-inflammatory effects due to its important contents including oleic acids, phenolic acids, secoiridoids and flavonoids. The oral application of olive oil has been shown to have protective anti-inflammatory effects and accelerated epithelial healing.
  Interventions: Procedure: Virgin olive oil

INTERVENTIONS:
Drug: Chlorhexidine Gluconate 0.12 % Mouthwash + benzydamine hydrochloride — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Other Names: Kloroben Oral Rinse
  Arms: chlorhexidine gluconate plus benzydamine hydrochloride
Procedure: St. John's wort oil — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: St. John's wort oil
Procedure: Virgin olive oil — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Virgin olive oil

SUMMARY:
Surgical removal of impacted third molars is one of the most frequent procedures carried out in the oral and maxillofacial surgery clinics. There are a varying range of postoperative complications including pain, edema and swelling. Antibiotics, analgesics and mouthwashes are usually prescribed for the treatment of these complications. Patients undergoing impacted third molar surgery are frequently prescribed chlorhexidine mouthwashes with/without benzydamine hydrochloride. However, to preclude the adverse effects of these chemical agents, there has been a search for plant-derived alternatives with anti-inflammatory, antibacterial and analgesic properties as part of the oral care routine following surgical removal of impacted third molars. However, there is no study investigating the comparison of different essential oils in the literature. Thus, this multicenter study was aimed to evaluate the effects of St. John's wort oil and virgin olive oil on the postoperative complications and compared with chlorhexidine gluconate plus benzydamine hydrochloride mouthwash after the removal of impacted wisdom teeth.This study was aimed to evaluate the effects of St. John's wort oil, virgin olive oil, and chlorhexidine gluconate plus benzydamine hydrochloride on the postoperative complications after the removal of impacted wisdom teeth.

ELIGIBILITY:
Inclusion Criteria:

* be 18-40 years old
* has unilateral mandibular impacted third molars with similar angulation position according to Winter's classification (mesio-angular) and similar impaction degree according to Pell & Gregory's classification (class II, Level B).
* absence of any systemic disease
* absence of pregnancy/lactating state,

Exclusion Criteria:

* Patients with smoking habits, drug abuse, history of pericoronitis associated with the lower third molar
* not regularly coming to the controls

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serap KESKIN TUNC, PhD, Study Chair — Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tusba, Turkey, 65080
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine Gluconate Plus Benzydamine Hydrochloride: Chlorhexidine is one of the most commonly used medications after tooth extraction. It exhibits a wide spectrum of antiseptic, bactericidal and bacteriostatic effects. The most common side effect of chlorhexidine is oral discoloration, taste changes and allergic responses. Furthermore, it has been reported that chlorhexidine has cytotoxic effect on gingival fibroblasts, epithelial cells, neutrophils and red blood cells; also shows incremental trend in genotoxicity as the duration of usage is increased. Benzydamine hydrochloride is a nonsteroidal anti-inflammatory drug that elicits anti-inflammatory, analgesic, anesthetic and antimicrobial effects. It is often used in addition to the topical application of chlorhexidine.. However, side effects such as urticaria, erythema, pruritus, photosensitivity, bronchospasm and renal problems can be observed associated with the use of benzydamine. Patients were also instructed to rinse their mouth with 15 ml of chlorhexidine gluconate plus benzydamine for 30 s, 3 times a day, and continue until the 7th postoperative day.
- St. John's Wort Oil: St. John's Wort (Hypericum perforatum) is a European medicinal plant with a history of more than 2000 years which possessing a variety of important constituents including phloroglucinols (hyperforin and adhyperforin), naphthodianthrones (hypericin and pseudohypericin), xanthones, essential oil, biflavones (biapigenin and amentoflavone), flavonol derivatives and phenolic compounds. The important components of St. John's Wort such as hypericin and hyperforin exert anti-inflammatory, antimicrobial, anticancer effects as well as stimulating tissue growth and differentiation. Hypericin exhibits anti-inflammatory effects by inhibiting the production of interleukin-12; whereas hyperforin reveals this effect by inhibiting the mechanisms of cyclooxygenase 1, 5-lipoxygenase and prostaglandin E2. St. John's Wort oil is extracted by maceration of the hypericum herb in carrier oil, such as virgin olive oil. Patients were also instructed to rinse their mouth with 15 ml of St. John's oil for 30 s, 3 times a day, and continue until the 7th postoperative day.
- Virgin Olive Oil: The olive oil, a product extracted from the fruit of Olea europaea, exerts also antioxidant and anti-inflammatory effects due to its important contents including oleic acids, phenolic acids, secoiridoids and flavonoids. The oral application of olive oil has been shown to have protective anti-inflammatory effects and accelerated epithelial healing. Patients were also instructed to rinse their mouth with 15 ml of virgin olive oil for 30 s, 3 times a day, and continue until the 7th postoperative day.
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Started | 30 | 30 | 30
Completed | 26 | 26 | 29
Not Completed | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Eighty-one healthy individuals who were in need of having impacted third molar surgery between August 2018 and March 2019 were included in this study. The inclusion criteria were being 18-40 years old, have asymptomatic unilateral mandibular impacted third molars with similar angulation positions according to Winter's classification (mesioangular), and having a similar impaction degree according to Pell and Gregory's classification (class II, level B).
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil | Total
Number analyzed (Participants) | 26 | 26 | 29 | 81
Age, Categorical [Count of Participants; unit: Participants] — Population: Total of 90 patients met the inclusion criteria; however, 9 patients were excluded from the study as they did not attend at least one follow-up appointment during the study period.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 26 | 26 | 29 | 81
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total of 90 patients met the inclusion criteria; however, 9 patients were excluded from the study as they did not attend at least one follow-up appointment during the study period.
  Participants
    Female | 19 | 21 | 23 | 63
    Male | 7 | 5 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: To record the level of pain, patients were instructed to rate it on a 100-mm visual analog scale (VAS) was used wherein 0 indicated no pain and 100 indicated the worst pain imaginable.
Time Frame: Postoperatif 1st day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 51.4 (21.9) | 56.3 (24.1) | 60.9 (25.1)

2. Primary Outcome: Postoperative Jaw Function
Description: For the assessment of difficulty during jaw function, patients were asked to rate it on a 100-mm VAS, wherein 0 indicated no limitation and 100 indicated severe limitation.
Time Frame: Postoperatif 1st day
Population: The inclusion criteria were being 18-40 years old, ave asymptomatic unilateral mandibular impacted third molars with similar angulation positions according to Winter's classification (mesioangular), and having similar impaction degree according to Pell and Gregory's classification (class II, level B). Patients with smoking habits, drug abuse, and history of pericoronitis associated with the lower third molar were excluded from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 61.5 (23.6) | 63.9 (24.7) | 65.9 (25.6)

3. Primary Outcome: Postoperative Swelling
Description: Facial swelling was assessed using a thread and millimeter ruler and averaged the following five measurements: Distance I (from the angle of the mandible to labial commissure); Distance II (from the angle of the mandible to the nasal border); Distance III (from the angle of the mandible to the external corner of the eye); Distance IV (from the angle of the mandible to tragus) and Distance V (from the angle of the mandible to soft pogonion). For evaluation of changes in the abovementioned distances during the postoperative period, the percentage of facial swelling was calculated by subtracting the preoperative measurements from the postoperative measurements then divided by the preoperative measurements and multiplied by 100.
Time Frame: Postoperative 1st day
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
percent change | 4.93 (7.60) | 3.90 (5.66) | 4.96 (5.37)

4. Primary Outcome: Postoperative Trismus
Description: For evaluation of trismus, the percentage of difference in maximum mouth opening during the postoperative period (B) was calculated by subtracting the preoperative measurement (A) from the postoperative measurement then dividing by the preoperative measurement (A) and multiplying by 100 (percentage of difference = [B - A]/B × 100).
Time Frame: Postoperative 1st day
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
percent change | 30.1 (8.7) | 28.7 (9.7) | 28.1 (7.8)

5. Primary Outcome: Postoperative Pain
Description: To record the level of pain, patients were instructed to rate it on a 100-mm visual analog scales (VAS) was used wherein 0 indicated no pain and 100 indicated the worst pain imaginable.
Time Frame: Postoperatif 2nd day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 44.5 (25.4) | 44.1 (23.4) | 55.8 (25.6)

6. Primary Outcome: Postoperative Jaw Function
Description: as for outcome 2
Time Frame: Postoperatif 2nd day
Population: The inclusion criteria were being 18-40 years old, have asymptomatic unilateral mandibular impacted third molars with similar angulation positions according to Winter's classification (mesioangular), and having similar impaction degree according to Pell and Gregory's classification (class II, level B).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 55.8 (25.4) | 51.9 (25.1) | 62.0 (25.1)

7. Primary Outcome: Postoperative Pain
Description: as for outcome 5
Time Frame: Postoperatif 3rd day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 36.2 (28.7) | 31.6 (22.6) | 40.6 (21.9)

8. Primary Outcome: Postoperative Jaw Function
Description: as for outcome 2
Time Frame: Postoperatif 3rd day
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 47.8 (28.1) | 42.5 (24.5) | 47.2 (20.5)

9. Primary Outcome: Postoperative Swelling
Description: as for outcome 3
Time Frame: Postoperative 3rd day
Measure: Mean (Standard Deviation); unit: percentage of swelling
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
percentage of swelling | 4.09 (7.18) | 3.24 (4.88) | 4.22 (4.43)

10. Primary Outcome: Postoperative Trismus
Description: as for outcome 4
Time Frame: Postoperative 3rd day
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
percent change | 33.8 (8.7) | 32.4 (9.1) | 31.6 (6.7)

11. Primary Outcome: Postoperative Pain
Description: as for outcome 5
Time Frame: Postoperatif 4th day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 33.6 (27.7) | 30.3 (22.4) | 30.4 (9.2)

12. Primary Outcome: Postoperative Jaw Function
Description: as for outcome 2
Time Frame: Postoperatif 4th day
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 44.4 (25.3) | 36.6 (22.5) | 35.1 (20.4)

13. Primary Outcome: Postoperative Pain
Description: as for outcome 5
Time Frame: Postoperatif 5th day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 22.0 (23.7) | 17.7 (16.0) | 26.3 (23.6)

14. Primary Outcome: Postoperative Jaw Function
Description: as for outcome 2
Time Frame: Postoperatif 5th day
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 29.5 (19.8) | 26.1 (20.1) | 28.6 (21.7)

15. Primary Outcome: Postoperative Pain
Description: as for outcome 5
Time Frame: Postoperatif 6th day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 16.3 (16.8) | 15.5 (18.6) | 19.0 (17.6)

16. Primary Outcome: Postoperative Jaw Function
Description: as for outcome 2
Time Frame: Postoperatif 6th day
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 19.5 (14.9) | 21.4 (19.1) | 20.6 (17.6)

17. Primary Outcome: Postoperative Pain
Description: as for outcome 5
Time Frame: Postoperatif 7th day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 10.5 (15.5) | 10.7 (18.5) | 9.6 (11.2)

18. Primary Outcome: Postoperative Jaw Function
Description: as for outcome 2
Time Frame: Postoperatif 7th day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
score on a scale | 11.5 (11.0) | 13.9 (18.0) | 13.8 (15.4)

19. Primary Outcome: Postoperative Swelling
Description: as for outcome 3
Time Frame: Postoperative 7th day
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
percent change | 2.66 (7.13) | 1.58 (4.22) | 2.30 (3.65)

20. Primary Outcome: Postoperative Trismus
Description: as for outcome 4
Time Frame: Postoperative 7th day
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
Number analyzed (Participants) | 26 | 26 | 29
percent change | 38.7 (6.8) | 38.3 (8.3) | 36.7 (8.7)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Chlorhexidine Gluconate Plus Benzydamine Hydrochloride | St. John's Wort Oil | Virgin Olive Oil
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/29

LIMITATIONS AND CAVEATS:
The limitation of this study is the lack of microbiological evaluation which might ascertain the antibacterial efficacy of these essential oils in oral surgical procedures. Thus, for future prospects, it would be enlightening to increase the number of studies to investigate other secondary variables including microbiological assessment, different types of administration, and as well as cost-effectiveness of these plant-derived agents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04373421/Prot_SAP_000.pdf